CLINICAL TRIAL: NCT00002898
Title: MMT 95 Study For Rhabdomyosarcoma and Other Malignant Soft Tissue Tumors of Childhood
Brief Title: Surgery Followed by Chemotherapy in Treating Young Patients With Soft Tissue Sarcoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Societe Internationale d'Oncologie Pediatrique (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000065228; SIOP-MMT-95; EU-96035
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 1999-05

CONDITIONS: Childhood Malignant Fibrous Histiocytoma of Bone; Sarcoma
Keywords: embryonal childhood rhabdomyosarcoma; alveolar childhood rhabdomyosarcoma; pleomorphic childhood rhabdomyosarcoma; mixed childhood rhabdomyosarcoma; embryonal-botryoid childhood rhabdomyosarcoma; nonmetastatic childhood soft tissue sarcoma; childhood fibrosarcoma; childhood synovial sarcoma; childhood malignant hemangiopericytoma; childhood liposarcoma; childhood alveolar soft-part sarcoma; childhood leiomyosarcoma; childhood neurofibrosarcoma; childhood angiosarcoma; childhood epithelioid sarcoma; childhood malignant fibrous histiocytoma of bone; childhood malignant mesenchymoma; previously untreated childhood rhabdomyosarcoma; childhood desmoplastic small round cell tumor; localized Ewing sarcoma/peripheral primitive neuroectodermal tumor
MeSH Terms: conditions — Sarcoma; Fibrosarcoma; Hemangiopericytoma, Malignant; Liposarcoma; Hemangiosarcoma; Malignant mesenchymal tumor; Desmoplastic Small Round Cell Tumor; Neuroectodermal Tumors, Primitive, Peripheral | interventions — Dactinomycin; Carboplatin; Cyclophosphamide; Epirubicin; Etoposide; Ifosfamide; Vincristine; Chemotherapy, Adjuvant; Neoadjuvant Therapy; Brachytherapy; Radiotherapy

INTERVENTIONS:
Biological: dactinomycin
Drug: carboplatin
Drug: cyclophosphamide
Drug: epirubicin hydrochloride
Drug: etoposide
Drug: ifosfamide
Drug: vincristine sulfate
Procedure: adjuvant therapy
Procedure: conventional surgery
Procedure: neoadjuvant therapy
Radiation: brachytherapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one chemotherapy drug with surgery and/or radiation therapy may kill more tumor cells.

PURPOSE: This randomized phase III trial is studying surgery followed by different regimens of combination chemotherapy given together with radiation therapy and/or additional surgery to compare how well they work in treating patients with soft tissue sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess whether good survival rates can be maintained for patients with stage I (pathologic T1) soft tissue sarcomas (STS) treated with limited chemotherapy after complete surgical resection, and whether disease-free survival can be improved by improving the precision of pretreatment staging and the assessment of the completeness of the resection.
* Compare the survival of patients with high-risk nonmetastatic STS treated with alternating regimens of carboplatin, epirubicin, and vincristine (CEV) and ifosfamide, vincristine, and etoposide (IVE) vs continuation of ifosfamide, vincristine, and dactinomycin (IVA) after initial therapy with IVA.
* Assess whether the improved outcome seen for patients with stage III (node positive) STS in an earlier protocol (SIOP-MMT-89) can be maintained with 3 courses of alternating CEV/IVE without altering local therapy.
* Compare outcome of patients with nonmetastatic STS to those with stage IV STS who are registered on this protocol but referred to treatment on the European Intergroup Stage IV Study.
* Assess survival and the risk of late sequelae in patients with non-rhabdomyosarcoma malignant mesenchymal tumors treated on this protocol.
* Evaluate the role of neoadjuvant chemotherapy, new prognostic factors (e.g., ploidy, histologic grading), and recommendations for the management of fibrosarcoma in infants and of fibromatoses.
* Assess ifosfamide nephrotoxicity based on total dose administered and the long-term toxicity based on the potential predictive value of early evidence of nephrotoxicity.

OUTLINE: This is a randomized study for patients with high-risk, nonmetastatic sarcoma, except those with the following characteristics: age less than 6 months, stage I/II non-alveolar orbital tumor, stage III disease, or age less than 3 years with parameningeal disease. Patients are stratified according to disease type (rhabdomyosarcoma (RMS) vs non-RMS disease), parameningeal site of disease, and participating center. Patients with RMS are further randomized by alveolar histology. Randomization occurs after the first course of chemotherapy.

All patients, regardless of disease stage, are registered to this study and outcome is followed, although patients with metastatic RMS or non-RMS malignant mesenchymal tumors are referred for treatment on the SIOP-MMT-98 study. Patients diagnosed more than 8 weeks prior to entry or who are unavailable for follow-up are not treated on study. Doses are modified for patients under 1 year of age or under 10 kg of body weight. All other patients are assigned therapy based on risk group.

After surgery, patients with complete resection and with proven or possible chemosensitive histologies proceed to chemotherapy on the low-risk regimen. Patients with questionable completeness of resection proceed to chemotherapy for standard-risk or high-risk tumors, as appropriate. Regardless of resection results, patients who underwent scrotal surgery for paratesticular tumors proceed to chemotherapy for standard-risk tumors. Alveolar RMS is considered high risk.

LOW-RISK TUMORS (T1 N0 M0): Strategy 951

* Tumors must be resectable without extensive, mutilating surgery, and resection margins must be microscopically negative at all sites. Patients with positive margins may undergo re-excision.
* Vincristine is administered weekly for 4 weeks with dactinomycin given on the same day as the first and fourth doses of vincristine. The course is repeated once after a 3-week rest.

STANDARD-RISK TUMORS (T1-2 N0 M0): Strategy 952

* After resection as above, patients with incompletely resected T1 tumors, completely resected T1 tumors that extended beyond the tissue or organ of origin, or completely or incompletely resected T2 tumors at favorable sites (vagina, uterus, or paratesticular region) receive chemotherapy on this regimen.
* Ifosfamide, vincristine, and dactinomycin (IVA) is started within 8 weeks of surgery and administered every 3 weeks for 3 courses; during this course only, vincristine is administered weekly throughout the 6 weeks. Response is assessed at week 8.
* Patients with at least a 50% response at week 8 receive 3 more courses of IVA and are reassessed at week 17; those with a complete response (CR) discontinue treatment, while those with less than a CR begin local therapy (described below) on week 18 concurrently with 3 more courses of IVA (unless no further response was seen after week 8).
* Patients with less than a 50% response at week 8 receive carboplatin, epirubicin, and vincristine (CEV) on weeks 9, 15, and 21 and ifosfamide, vincristine, and etoposide (IVE) on weeks 12, 18, and 24. Patients with less than a CR at week 17 receive concurrent local therapy beginning at week 18.

HIGH-RISK TUMORS: Strategy 953

* Patients with high-risk tumors after surgery are randomized to IVA as in strategy 952 (Arm I) or to 3 weeks of IVA (1 course) as in Strategy 952 followed by CEV and IVE as in Strategy 952 (Arm II). Response is assessed at week 8. Patients with parameningeal disease who are at least 3 years of age proceed to radiotherapy at week 9, regardless of response.
* Patients on Arm I with at least a 50% response at week 8 receive 3 more courses of IVA and are reassessed at week 17; those who continue to respond between weeks 8 and 17 receive 3 additional courses of IVA. Patients with no further response receive 4 alternating courses of CEV and IVE. All patients with less than a CR at week 17 begin local therapy on week 18 concurrently with the additional chemotherapy. Patients on Arm I with less than a 50% response at week 8 receive alternating CEV and IVE as in Strategy 952. Patients with less than a CR at week 17 begin concurrent local therapy at week 18.
* Patients on Arm II who have at least a 50% response at week 8 continue treatment with 2 courses of sequential IVA, CEV, and IVE. Local therapy is concurrently administered, beginning on week 18, to patients who have not achieved a CR by week 17. Patients on Arm II who have less than a 50% response at week 8 proceed immediately to local therapy with additional chemotherapy at the investigator's discretion. Patients with less than a CR after local therapy are considered for treatment on a phase II protocol.

LOCAL THERAPY

* Local therapy consists of conservative resection of residual disease (unless more debilitating surgery is appropriate). Patients with residual disease after surgery undergo external-beam radiotherapy 5 days per week for 6-7 weeks or brachytherapy; hyperfractionation is specifically excluded. For patients receiving radiotherapy, the dactinomycin dose in the IVA regimen is omitted from the middle course of chemotherapy and possibly the last course of chemotherapy during concurrent administration. Patients receiving alternating CEV and IVE have the courses reversed during concurrent radiotherapy, with possible omission of epirubicin for the third course.
* Radical surgery is considered for any patient who has residual disease at week 27.

TREATMENT FOR RELAPSE

* Patients treated with Strategy 951 proceed to therapy with at least 6 alternating courses of IVE and CEV, with local therapy initiated after the second course. Other patients receive at least 6 alternating courses of CEV and vincristine, carboplatin, and etoposide (modified Vincaepi), with local therapy initiated after the second course. Patients who have already received either regimen may be re-treated with carboplatin and etoposide and vincristine and cyclophosphamide if relapse occurs more than 6 months after treatment, while those who relapse in less than 6 months are considered for phase II chemotherapy trials. Patients with metastatic relapse are evaluated for bone marrow or peripheral blood stem cell transplantation.

Patients are followed every 2 months until 2 years after diagnosis, every 3 months for 1 year, every 6 months for 2 years, and then annually until 10 years after diagnosis.

PROJECTED ACCRUAL: A total of 400 patients with high-risk nonmetastatic disease will be accrued for this study within approximately 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary soft tissue sarcoma:

  * Rhabdomyosarcoma
  * Non-rhabdomyosarcoma
  * Soft tissue primitive neuroectodermal tumor (PNET)
  * Extraosseous Ewing's sarcoma

PATIENT CHARACTERISTICS:

Age:

* Under 18

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

PRIOR CONCURRENT THERAPY:

Biologic:

* Not specified

Chemotherapy:

* Not specified

Endocrine:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Prior primary surgery allowed

Other:

* No other prior therapy

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 400 (Estimated)
Dates: Start 1995-01; Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M. C. G. Stevens, MD, Study Chair — Institute of Child Health at University of Bristol
Locations (1):
- Institute of Child Health, Bristol, England, United Kingdom

REFERENCES:
- [Background] Chisholm JC, Marandet J, Rey A, Scopinaro M, de Toledo JS, Merks JH, O'Meara A, Stevens MC, Oberlin O. Prognostic factors after relapse in nonmetastatic rhabdomyosarcoma: a nomogram to better define patients who can be salvaged with further therapy. J Clin Oncol. 2011 Apr 1;29(10):1319-25. doi: 10.1200/JCO.2010.32.1984. Epub 2011 Feb 28. PMID 21357778
- [Background] Orbach D, Mc Dowell H, Rey A, Bouvet N, Kelsey A, Stevens MC. Sparing strategy does not compromise prognosis in pediatric localized synovial sarcoma: experience of the International Society of Pediatric Oncology, Malignant Mesenchymal Tumors (SIOP-MMT) Working Group. Pediatr Blood Cancer. 2011 Dec 15;57(7):1130-6. doi: 10.1002/pbc.23138. Epub 2011 Apr 14. PMID 21495161
- [Background] Defachelles AS, Rey A, Oberlin O, Spooner D, Stevens MC. Treatment of nonmetastatic cranial parameningeal rhabdomyosarcoma in children younger than 3 years old: results from international society of pediatric oncology studies MMT 89 and 95. J Clin Oncol. 2009 Mar 10;27(8):1310-5. doi: 10.1200/JCO.2008.19.5701. Epub 2009 Feb 9. PMID 19204197
- [Result] Oberlin O, Rey A, Sanchez de Toledo J, Martelli H, Jenney ME, Scopinaro M, Bergeron C, Merks JH, Bouvet N, Ellershaw C, Kelsey A, Spooner D, Stevens MC. Randomized comparison of intensified six-drug versus standard three-drug chemotherapy for high-risk nonmetastatic rhabdomyosarcoma and other chemotherapy-sensitive childhood soft tissue sarcomas: long-term results from the International Society of Pediatric Oncology MMT95 study. J Clin Oncol. 2012 Jul 10;30(20):2457-65. doi: 10.1200/JCO.2011.40.3287. Epub 2012 Jun 4. PMID 22665534